CLINICAL TRIAL: NCT03633578
Title: Relationship Between Complexity and Pain in a Walking Task With Distraction in the Chronic Low Back Pain Patient by Fractal Analysis: Pilot Study
Brief Title: Complexity & Distraction in LBP
Acronym: CoDiLoBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LOCAL/2017/AH-01; 2017-A02839-44 (Other: ANSM)
Record Dates: First submitted 2018-08-14; First posted 2018-08-16 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2020-12

CONDITIONS: Chronic Low Back Pain; Gait; Motor Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional group (Experimental): Patients are asked to walk ont a treadmill in four conditions: with and without distraction (virtual environment) and at different speed (comfortable vs high).
  Interventions: Behavioral: walk test

INTERVENTIONS:
Behavioral: walk test — The patient will have to walk on a treadmill in four different conditions:
  * without distraction at preferential speed
  * with distraction at preferential speed
  * without distraction at the speed of 130% of the preferential speed
  * with distraction at the speed of 130% of the preferential speed

SUMMARY:
Motor control, notably expressed through the complexity of the variability of the locomotor pattern, is disturbed at the central level by an apprehension of pain and movement, more than pain itself (or by biomechanical / structural damage of the spine) in chronic low back pain (cLBP) patients.

The aim of this study is to control that variability is reduced during gait at comfortable level and to test that distraction can reduce pain avoidance and therefore increase variability in cLBP patients.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have his informed consent and signed the consent form.
* The patient must be affiliated or beneficiary of a health insurance plan
* The patient is at least 18 years old and under 75 years old
* Patients with common chronic low back pain for more than 6 months

Exclusion Criteria:

* The subject participates in another interventional study
* The subject is in an exclusion period determined by a previous study
* The subject is under the protection of justice, guardianship or curatorship
* The subject refuses to sign the consent
* It is impossible to inform the subject
* Chronic symptomatic low back pain (tumoral pathology, infectious, or progressive inflammatory)
* Unable to walk for more than 10 minutes (during interrogation)
* Lower limb pain (EVA lower limb (s) ≥ Lumbar EVA)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-05-17 (Actual); Study Completion 2018-05-17 (Actual)

PRIMARY OUTCOMES:
Estimation of the fractal exponent when walking without distraction at preferential speed | Day 0
  [0,5; 1,5]
Estimation of the fractal exponent when walking with distraction at preferential speed | Day 0
  [0,5; 1,5]
Estimation of the fractal exponent when walking without distraction at the speed of 130% of the preferential speed | Day 0
  [0,5; 1,5]
Estimation of the fractal exponent when walking with distraction at the speed of 130% of the preferential speed | Day 0
  [0,5; 1,5]

SECONDARY OUTCOMES:
EVA after walking without distraction at preferential speed | Day 0
  [0; 100]
EVA after walking with distraction at preferential speed | Day 0
  [0; 100]
EVA after walking without distraction at the speed of 130% of the preferential speed | Day 0
  [0; 100]
EVA after walking with distraction at the speed of 130% of the preferential speed | Day 0
  [0; 100]
Reaction time to auditory stimuli without distraction at preferential speed | Day 0
  second
Reaction time to auditory stimuli with distraction at preferential speed | Day 0
  second
Reaction time to auditory stimuli without distraction at the speed of 130% of the preferential speed | Day 0
  second
Reaction time to auditory stimuli with distraction at the speed of 130% of the preferential speed | Day 0
  second
Tampa Scale for kinesophobia | Day 0
  The total score ranges between 17 and 68. A high value on the Tampa Scale for the "Tampa Scale for kinesophobia" indicates a high degree of kinesiophobia
Dallas Pain Questionnaire for Back Pain | Day 0
  This questionnaire has been designed to give health care provider information as to how pain affects daily activities. It assesses the impact of low back pain (LBP) on four components (daily activities, work and leisure activities, anxiety/depression, and social interest) (expressed as a value between 0 and 100) of daily life.The higher the score, the more the low back pain has an impact on the quality of life.
Quebec Back Pain Disability Index | Day 0
  The item scores were summed for a total score between 0 and 100, with higher numbers representing greater levels of disability.
Fear Avoidance Belief Questionnaire (FABQ) | Day 0
  The Fear Avoidance Belief Questionnaire is a two-part questionnaire assessing fear, avoidance, and beliefs about professional activity and physical activity.
  The FABQ physical activity score of 14 responds better to a cognitive/behavioral approach and de-emphasize the traditional pain specific treatment goals. The "Fear Avoidance Belief Questionnaire" Work score that is >18 has a decrease likelihood of success from a joint manipulation/mobilization treatment approach. The "Fear Avoidance Belief Questionnaire" Work score of 34 or greater increases the risk for prolonged disability and will most likely require a multi-disciplinary approach to treatment.
Hospital and Anxiety Depression Scale | Day 0
  Score:
  0-7 = Normal 8-10 = Borderline abnormal (borderline case) 11-21 = Abnormal (case)

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Dupeyron, Pr, Principal Investigator — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- Nimes University Hospital, Nîmes, France

REFERENCES:
- [Result] Homs AF, Dupeyron A, Torre K. Relationship between gait complexity and pain attention in chronic low back pain. Pain. 2022 Jan 1;163(1):e31-e39. doi: 10.1097/j.pain.0000000000002303. PMID 34001770